CLINICAL TRIAL: NCT07404852
Title: Neuromodulation Using Vagus Nerve Stimulation Following Ischemic Stroke as Therapeutic Adjunct 2
Brief Title: Non-invasive Vagus Nerve Stimulation to Reduce Inflammation and Brain Injury Blood Biomarkers Following an Acute Ischemic Stroke
Acronym: NUVISTA 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Osvaldo J. Laurido-Soto, MD, Assistant Professor of Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 202601166
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Large Vessel Occlusion; Acute Ischemic Stroke
Keywords: Acute ischemic stroke; large vessel occlusion; cytokines; vagus nerve stimulator; brain injury biomarkers
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This is a randomized open-label, with blinded outcome pilot study to evaluate the effect on inflammatory and brain injury laboratory values and explore clinical outcomes in patients who present with ischemic strokes due to large vessel occlusions and are treated with either current accepted management, or accepted management in addition to transcutaneous auricular vagus nerve stimulation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients enrolled in the trial will be randomized to treatment with electrical stimulation to the auricular branch of the vagus nerve (intervention) or no stimulation to the auricular branch of the vagus nerve (Sham) via an auricular, transcutaneous vagus nerve stimulator. All patients will be fitted with the device, the investigators will attach the electrodes to the left ear. Patients are blinded to the intervention and study personnel will be unblinded, except those performing the laboratory testing and result analyses. Care provider team will be blinded to which treatment group the patient is on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment - Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator (Experimental): All patients will be fitted with the device, the investigator will attach an electrode to the left ear. Stimulation sessions will occur for 20 minutes twice daily during the inpatient period, the investigator will stimulate the auricular branch of the vagus nerve. Patients' will be treated with the following parameters: frequency 20 Hz, pulse width 250 μm, and and a fixed intensity of 0.5 milliampere.
  Interventions: Device: transcutaneous auricular vagal nerve stimulation
- Control - No Stimulation Transcutaneous Auricular Vagal Nerve Stimulator (Sham Comparator): All patients will be fitted with the device, the investigator will attach an electrode to the left ear. Sham stimulation sessions will occur for 20 minutes twice daily during the inpatient period. Patients assigned to the controls arm will have no electricity applied to the auricular branch of the vagus nerve.
  Interventions: Device: Sham transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagal nerve stimulation — Stimulus of the auricular branch of the vagal nerve with the transcutaneous auricular vagal nerve stimulation.
  Arms: Treatment - Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator
Device: Sham transcutaneous vagal nerve stimulation — Patients assigned to the controls arm will have no electricity applied to the Auricular Branch of the Vagus Nerve.
  Arms: Control - No Stimulation Transcutaneous Auricular Vagal Nerve Stimulator

SUMMARY:
This is a randomized open-label, with blinded outcome pilot study to evaluate the effect on inflammatory and brain injury laboratory values and explore clinical outcomes in patients who present with ischemic strokes due to large vessel occlusions and are treated with either current accepted management, or accepted management in addition to transcutaneous auricular vagal nerve stimulation.

DETAILED DESCRIPTION:
Ischemic stroke is a leading cause of death and long-term disability worldwide. Large vessel occlusion (LVO) accounts for ~38% of acute ischemic strokes (AIS) and is associated with disproportionately poor outcomes: without treatment, 64% of patients are dead or dependent at six months, and even after successful mechanical thrombectomy, nearly half have poor functional recovery. These data highlight a critical unmet need for adjunctive therapies that limit secondary brain injury following reperfusion.

Neuroinflammation is a major contributor to ischemic brain injury and neurologic deterioration after AIS. In experimental models, inhibition of inflammatory pathways reduces infarct size and improves outcomes, and in human AIS, elevations in pro-inflammatory cytokines are associated with worse recovery. However, clinical trials targeting individual inflammatory mediators have failed, suggesting that effective therapy may require coordinated modulation of multiple immune pathways rather than blockade of a single target. Vagus nerve stimulation (VNS) engages an evolutionary conserved neuroimmune reflex that broadly regulates innate and adaptive immune responses. While implantable VNS is not feasible in acute stroke, non-invasive transauricular VNS (taVNS) enables rapid deployment in emergent settings.

We recently completed the Neuromodulation Using Vagus Nerve Stimulation Following Ischemic Stroke as Therapeutic Adjunct (NUVISTA) pilot randomized trial (n=35) in AIS patients with LVO. taVNS was rapidly deployable and safe, significantly attenuated the trajectory of plasma interleukin-6 (IL-6) and other inflammatory mediators, and demonstrated encouraging signals of improved clinical outcomes. These findings support further mechanistic and translational investigation in a well-powered cohort.

The central hypothesis of this proposal is that taVNS engages endogenous neuroimmune reflexes to reprogram peripheral immune responses following LVO AIS, resulting in reduced systemic inflammation, attenuation of neuroaxonal injury, and improved early recovery. We will test this hypothesis in a randomized, sham-controlled clinical study of 65 AIS patients

Patients enrolled in the trial will be randomized to treatment with electrical stimulation to the auricular branch of the vagus nerve (intervention) or no stimulation to the auricular branch (Sham) via an auricular, transcutaneous vagus nerve stimulator. All patients will be fitted with the device, the investigators will attach the ear electrodes to the left ear. Stimulation sessions will occur for 20 minutes twice daily during the inpatient period. Patients will have electricity applied to the different nerves depending on the randomization, they will be treated with stimulation with the following parameters: frequency 20 Hz, pulse width 250 μm, and a fixed intensity of 0.5 milliampere. The amplitude of stimulation may be reduced if a patient complains of discomfort at the site of stimulation. The site of stimulation will be inspected daily before and after treatment to ensure there is no redness or irritation at the site. The investigators will obtain laboratory samples on admission, day 0, and every 1.5 days till day 7 or discharge (whichever occurs first) to assess the patients inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who present with acute ischemic strokes due to large vessel occlusions

Exclusion Criteria:

* <18 years old
* patients with presumed chronic large vessel occlusions
* NIHSS<6
* pre-morbid modified Rankin score (mRS) >2
* unable to initiate treatment under 24 hours from symptom discovery
* Chronic or acute infection, Recent surgery, active immune disease
* life expectancy <3 months
* patients' undergoing active cancer or immunosuppressive/modulating therapy
* patients with sustained bradycardia on arrival with a heart rate <50 beats per minute.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2027-11-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Brain Derived Tau | 7 days
  The primary endpoints of the study will include changes in the levels of brain injury biomarkers measured at onset and every 1.5 days till day 7, or discharge (whichever occurs first), this includes: Brain Derived Tau (BD-tau). The investigators will measure BD-tau in aliquots from the plasma with mononuclear antibodies that recognizes a protein of 48 to 68 kilodalton specific to BD-tau. A functional assay will be measured in picogram/milliliter. Will utilize a high sensitivity assays to minimize floor effects.
Neurofilament light chain | 7 days
  The primary endpoints of the study will include changes in the levels of brain injury biomarkers measured at onset and every 1.5 days till day 7, or discharge (whichever occurs first), this includes: Neurofilament light chain (NfL). The investigators will measure NfL in aliquots from the plasma with mononuclear antibodies that recognizes a protein of 68-70 kilodalton specific to NfL. A functional assay will be measured in picogram/milliliter. Will utilize a high sensitivity assays to minimize floor effects.
Interleukin - 1b - Changes and Differences in the Levels | 7 days
  The primary endpoints of the study will include changes in the levels of inflammatory markers measured at onset and every 1.5 days till day 7, or discharge (whichever occurs first), this includes: Interleukin (IL) -1b. The investigators will measure IL-1b in aliquots from the plasma with mononuclear antibodies that recognizes a protein of 17-31 kilodalton specific to IL-1b. A functional assay will be measured in picogram/milliliter. Will utilize a high sensitivity assays to minimize floor effects.
Interleukin - 6 - Changes and Differences in the Levels | 7 days
  The primary endpoints of the study will include changes in the levels of inflammatory markers measured at onset and every 1.5 days till day 7, or discharge (whichever occurs first), this includes: Interleukin (IL) - 6. The investigators will measure IL-6 in aliquots from the plasma with mononuclear antibodies that recognizes a protein of 26 kilodalton specific to IL-6. A functional assay will be measured in picogram/milliliter. Will utilize a high sensitivity assays to minimize floor effects.
Tumor Necrosis Factor Alpha - Changes and Differences in the Levels | 7 days
  The primary endpoints of the study will include changes in the levels of inflammatory markers measured at onset and every 1.5 days till day 7, or discharge (whichever occurs first), this includes: Tumor necrosis factor alpha (TNF-a). The investigators will measure IL-1b in aliquots from the plasma with mononuclear antibodies that recognizes a protein of 17 kilodalton specific to TNF-a. A functional assay will be measured in picogram/milliliter. Will utilize a high sensitivity assays to minimize floor effects.

SECONDARY OUTCOMES:
Change in NIH Stroke Scale (NIHSS) | 7 days
  This is a clinical secondary exploratory endpoints. The NIH Stroke Scale (NIHSS) is a clinical tool used to assess stroke severity, the score ranges from 0 up to 42 (higher is more severe). It will be assessed daily by the investigators and at time of discharge. The investigators will assess differences in NIHSS dependent of the intervention arm.
Modified Ranking Scale (mRS) | 90 days
  This is a clinical secondary exploratory endpoints. The Modified Ranking Scale (mRS) is a clinical tool used to assess functional status after suffering a stroke. It ranges from 0 up to 6. It will be assessed at day 90 over the phone. The investigators will assess differences in mRS dependent of the intervention arm.
  0 = no symptoms at all
  1. = No significant disability despite symptoms; able to carry out all usual duties and activities
  2. = Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance.
  3. = Moderate disability; requiring some help, but able to walk without assistance.
  4. = Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. = Severe disability; bedridden, incontinent and requiring constant nursing care and attention.
  6. = Dead

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient level data may be shared upon reasonable requested and approval by the institutions Human Research Protection Office
Time Frame: Once the trial is finished and publish. Estimated March 2028
Access Criteria: De-identified patient level data may be shared upon reasonable requested and approval by the institutions Human Research Protection Office

REFERENCES:
- [Background] Laurido-Soto OJ, Tan G, Nielsen SS, Huguenard AL, Donovan KM, Xu I, Giles J, Dhar R, Adeoye O, Lee JM, Leuthardt E. Transcutaneous Auricular Vagus Nerve Stimulation Reduces Inflammatory Biomarkers after Large Vessel Occlusion Stroke: Results of a Prospective Randomized Open-Label Blinded Endpoint Trial. Transl Stroke Res. 2025 Dec 22;17(1):7. doi: 10.1007/s12975-025-01405-6. PMID 41428140